CLINICAL TRIAL: NCT00098332
Title: A Phase I, Multi-Center, Open-Label, Safety and Pharmacokinetic, Repeat-Dose Study of Oral Forodesine Hydrochloride in Patients With Refractory Cutaneous T-Cell Lymphoma
Brief Title: Forodesine (BCX-1777) in Treating Patients With Refractory Stage IIA, Stage IIB, Stage III, Stage IVA, or Stage IVB Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: BIOCRYST-BCX1777-C-04-105; CDR0000405886 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2007-06

CONDITIONS: Lymphoma
Keywords: recurrent cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

INTERVENTIONS:
Drug: forodesine hydrochloride

SUMMARY:
RATIONALE: Forodesine (BCX-1777) may stop the growth of cancer cells by blocking the enzymes necessary for their growth.

PURPOSE: Phase I trial to study the effectiveness of BCX-1777 in treating patients who have refractory stage IIA, stage IIB, stage III, stage IVA, or stage IVB cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of forodesine (BCX-1777) in patients with refractory stage IIA-IVB cutaneous T-cell lymphoma.
* Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral forodesine (BCX-1777) once daily on days 1-28. Courses may be repeated in the absence of disease progression or unacceptable toxicity.

Patients are followed periodically.

PROJECTED ACCRUAL: Not specified.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous T-cell lymphoma

  * Refractory to prior treatment
  * Stage IIA, IIB, III, IVA, or IVB disease
* Measurable disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* AST and/or ALT ≤ 3 times upper limit of normal
* Hepatitis B and/or hepatitis C negative

Renal

* Creatinine clearance ≥ 40 mL/min

Immunologic

* Human T-cell lymphotrophic virus type I (HTLV-I) negative
* HIV negative
* No active serious infection not controlled by antibiotics

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known impaired absorption of the gastrointestinal tract
* No other illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 21 days since prior chemotherapy and recovered

Endocrine therapy

* Concurrent topical corticosteroids allowed provided patient remains on a stable dose

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior investigational agents and recovered
* No concurrent tanning bed use
* No other concurrent therapy for cutaneous T-cell lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama-Birmingham, Birmingham, Alabama
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Cancer and Blood Disease Center, Lecanto, Florida
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas